CLINICAL TRIAL: NCT06614114
Title: Albumin Bilirubin Index as a Predictor of Outcome of Variceal Bleeding
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba Sayed Zaki Bebe, Assiut, Assiut University
Other Study IDs: Alb/bl in variceal bleeding
Record Dates: First submitted 2024-09-09; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Prediction of Variceal Bleeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Albumin bilirubin index as a predictor of outcome of variceal bleeding

DETAILED DESCRIPTION:
This study is to clarify the predictive value of albumin bilirubin index for recurrent bleeding within 3 month after endoscopic treatment in patients with cirrhosis and EGVB

ELIGIBILITY:
Inclusion Criteria:

* age between 18-80 years old

Exclusion Criteria:

* Hcc Hematological disease

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients had developed variceal bleed and who had been admitted via emergency
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2024-09-24 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
prevelence of Variceal bleeding in high alb/bill index | 6 months
  Prevelence of bleeding in patient with cirrhosis

CONTACTS AND LOCATIONS:
Overall Officials: Heba Sayed Zaki, Principal Investigator — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Egypt